CLINICAL TRIAL: NCT06985849
Title: Effects of Feldenkrais and Otago Exercise Protocols for Mechanical Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0181
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feldenkrais method. (Experimental): Group A will receive awareness through movement lessons, which are verbally, guided explorations of movement, conducted by a physiotherapist. The Feldenkrais method intervention consisted of 10 structured lessons, each 30 minutes in duration, delivered twice weekly. The program aimed to enhance trunk mobility and overall function without pain. Lessons progressed sequentially, building upon previous sessions. Segment 1 (Lesson 1-2) focused on breathing awareness and trunk perception in supine position, gaining control of the pelvis, and freeing hip joints. Segment 2 (Lesson 3-4) addressed flexion-extension and self-care in supine and prone positions. Segment 3 (Lesson 5-6) targeted flexion-extension, rotation, and shoulder control. Segment 4 (Lesson 7-8) emphasized balance and walking. The final lessons (9-10) integrated previous themes, reinforcing functional improvement
  Interventions: Other: Feldenkrais method
- Otago exercise protocol. (Active Comparator): The study began by completing all 3-outcome measures by first asking about their pain intensity then by checking their balance through Berg Balance Scale and then checking the level of function through ODI questionere. The OEP included the following exercises: knee extension and knee flexion, hip abduction, calf raises, toe raises, sit to stand, semi squats from a standing position, tandem stand, tandem walk, sideways walking, backwards walking, heel walking, toe walking, one leg stand, and walking and turning around. All exercises will be performed with 10-20 repetitions, which will be progressed after 2 week
  Interventions: Other: Otago exercise protocol.

INTERVENTIONS:
Other: Feldenkrais method — "Activating flexors" "The pelvic clock"twisting)."Side lying lesson for improving the integration of arms, shoulders and spine" (reaching motion of shoulders in different directions)."Transitioning from supine to side lying to sitting" (lying supine involving flexion, extension, and twisting)."Twisting on the side" "Twisting from supine with head fixed to the side" (by limiting the movement of the head, the rib cage is forced to participate in the twisting motion) "Lengthening the hamstrings" "Arm circles" (lying on side, circling arms in different directions). "Rolling from supine to prone via hip rotation
  Arms: Feldenkrais method.
Other: Otago exercise protocol. — The study began by completing all 3-outcome measures by first asking about their pain intensity then by checking their balance through Berg Balance Scale and then checking the level of function through ODI questionere. The OEP included the following exercises: knee extension and knee flexion, hip abduction, calf raises, toe raises, sit to stand, semi squats from a standing position, tandem stand, tandem walk, sideways walking, backwards walking, heel walking, toe walking, one leg stand, and walking and turning around. All exercises will be performed with 10-20 repetitions, which will be progressed after 2 week.(12)
  Arms: Otago exercise protocol.

SUMMARY:
Low back pain (LBP) is a common health issue-affecting individual across diverse ages and socio- economic backgrounds, with approximately 80% of the population experiencing this musculoskeletal concern at some point in their lives. Despite its prevalence, the prognosis for LBP is generally favorable, emphasizing the importance of effective management strategies aimed at reducing pain and improving functional ability. The Feldenkrais Method and the Otago Exercise Programme (OEP) are two interdisciplinary approaches that have demonstrated promise in addressing mechanical non-specific low back pain. This study aims to evaluate the effectiveness of these two intervention protocols in alleviating chronic low back pain while concurrently enhancing functional abilities and reducing the risk of falls among older adults.

The study will be a randomized controlled trial conducted on participants. Data will be collected from Farooq hospital and Boston physiotherapy and wellness clinic. This study will be completed in time duration of 10 months after the approval of synopsis. Non-probability convenience sampling technique will be used and participant's age between 45-65, having mechanical low back pain for more than 3 months will be recruited in study after computer generated randomization. However, participants who have any chronic illness like recurrent spinal surgery, Malignancy, Spine Infection, Spinal fracture and congenital disturbance shall be excluded from this study. The subjects will be divided into two groups. Group A will receive awareness through movement sessions of trunk mobility, which will be guided verbally(such as rolling head left and right, bringing knees to chest, tilting to the sides, rolling pelvis.) and Group B will receive lower limb strength and balance exercises like knee extensions and hip abduction.

All these sessions will be of 30 minutes to for 2 sessions per week for 6 weeks. Pre and post assessments will be conducted and the tools that will be used are NPRS for pain, Universal goniometer for ROM, Functional disability (Oswestry Disability Index), Falls-related self-efficacy will be assessed by the Activities-Specific Balance Confidence (ABC) Scale. and Balance (Berg Balance Scale). Data will be analyzed by using SPSS version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* • Age group 18 to 65 year (3)

  * Both gender male and female
  * LBP (duration ≥ 3 months) (3)
  * NPRS score ≥ 4/10 (indicating moderate pain)
  * ODI: Score ≥ 20/100 (indicating moderate disability)
  * BBS: Score ≤ 45/56 (indicating balance impairment)
  * BC Scale score: ≤ 60/100 (indicating moderate to low balance confidence)
  * Ability to walk independently
  * No severe cognitive impairment
  * Patient willing to perform in the study

Exclusion Criteria:

* • Recurrent spinal surgery(3)

  * Malignancy
  * Spine Infection
  * Spinal fracture
  * Congenital disturbance
  * Severe LBP (NPRS ≥ 9/10)
  * Significant balance impairment (BBS ≤ 20/56)
  * Severe disability (ODI ≥ 60/100)
  * ABC Scale score: ≥ 80/100 (indicating high balance confidence)
  * Older individuals with specific health conditions, such as cardiovascular disease and diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale ( BBS) | baseline and fourth week
  It is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. Berg Balance Scale Sensitivity is 0.75-0.91 and Specificity is 0.67-0.85 (ability to identify those without balance impairment)It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Oswestry Disability Index (ODI) | baseline and fourth week
  It is a patient-completed questionnaire that gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. It was developed by Jeremy Fairbank and Graham Pynsent in Oswestry, England in 1980 and considered one of the best-accepted tools for assessment of low back pain. ODI Sensitivity (0.74-0.92) and Specificity is (0.63-0.85), The questionnaire examines the level of disability in 10 everyday activities of daily living. Each item consist of 6 statements which are scored from 0 to 5. With 0 indicating the least disability and 5 the greatest then the total score is calculated as a percentage, with 0% indicating no disability and 100% indicating the highest level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University
Locations (1):
- Farooq Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gianola S, Bargeri S, Del Castillo G, Corbetta D, Turolla A, Andreano A, Moja L, Castellini G. Effectiveness of treatments for acute and subacute mechanical non-specific low back pain: a systematic review with network meta-analysis. Br J Sports Med. 2022 Jan;56(1):41-50. doi: 10.1136/bjsports-2020-103596. Epub 2021 Apr 13. PMID 33849907
- [Background] Senbursa G, Pekyavas NO, Baltaci G. Comparison of Physiotherapy Approaches in Low Back Pain: A Randomized Controlled Trial. Korean J Fam Med. 2021 Mar;42(2):96-106. doi: 10.4082/kjfm.20.0025. Epub 2020 May 22. PMID 32438535
- [Background] Ahmadi H, Adib H, Selk-Ghaffari M, Shafizad M, Moradi S, Madani Z, Partovi G, Mahmoodi A. Comparison of the effects of the Feldenkrais method versus core stability exercise in the management of chronic low back pain: a randomised control trial. Clin Rehabil. 2020 Dec;34(12):1449-1457. doi: 10.1177/0269215520947069. Epub 2020 Jul 29. PMID 32723088